CLINICAL TRIAL: NCT06302244
Title: Multimodal Neuromonitoring in Patients With Severe Acute Brain Injury
Brief Title: Multimodal Neuromonitoring in Acute Brain Injury
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne-Sophie Worm Fenger, MD, PhD fellow, Rigshospitalet, Denmark
Other Study IDs: R-21075263
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Acute Brain Injury
Keywords: Brain injury; Intensive care; Neurointensive care; Anaesthesiology; Multimodal neuromonitoring
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Acute brain injury due to aneurysmal subarachnoid haemorrhage (SAH) or traumatic brain injury (TBI) is a condition with a high mortality, and surviving patients often have permanent disabilities. Multimodal neuromonitoring of intracranial pressure, brain tissue oxygen tension (PbtO2), and brain energy metabolism (measured with microdialysis (MD)) may help individualise the treatment of this patient group to protect the brain and potentially improve outcomes. However, there is still a significant lack of knowledge regarding the advantages and disadvantages of this type of monitoring.

The present study consists of four substudies with the overall aim of examining which factors are most influential for regulating commonly measured intracerebral parameters such as oxygenation, glucose, and lactate. Additionally, the influence of these of parameters on functional outcome and mortality will be explored.

The individual studies are detailed below:

DETAILED DESCRIPTION:
Substudy 1:

This study investigates the relationship between glucose in blood and microdialysate (MD-glucose) in patients with severe traumatic brain injury (TBI) or aneurysmal subarachnoid haemorrhage (SAH).

Substudy 2:

The aim of this substudy is to examine the contribution of arterial oxygen tension (PaO2) to PbtO2 in patients with acute brain injury. We hypothesize that there is an association between the two parameters, that this relationship is altered in patients with concurrent intracranial hypoertension, and that a higher burden of cerebral hypoxia is associated with poor functional outcome and mortality.

Substudy 3:

The study aims to estimate the contribution of systemic lactate to microdialysate lactate, hypothesizing that:

1. PbtO2 and cerebral perfusion pressure are independent predictors of microdialysate lactate in patients with cerebral hypoxia (PbtO2<20).
2. Systemic lactate is an independent predictor of microdialysis lactate in patients without cerebral hypoxia.

Substudy 4:

The study aims to establish whether there is a predictive threshold value of MD-glutamate for unfavourable functional outcome 6 months after ictus of brain injury. Additionally, we aim to explore whether there is a pattern of MD-glutamate that can predict episodes of neuroworsening.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the Neurointensive care unit at Rigshospitalet, Copenhagen
* Diagnosis of traumatic brain injury or subarachnoid haemorrhage
* Multimodal neuromonitoring consisting intracranial pressure, brain tissue oxygen tension, and/or cerebral microdialysis

Exclusion Criteria:

* Age below 18 years
* Acute brain injury due to causes other than the above mentioned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe acute brain injury and diagnosis of traumatic brain injury or subarachnoid haemorrhage admitted to the neurointensive care unit at Copenhagen University Hospital Rigshospitalet
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation between systemic glucose and microdialysis glucose | Throughout the duration of neuromonitoring in the neuro-ICU (1-30 days)
  Median goodness of fit (Pearsons R2)
Median goodness of fit (Pearsons R2) of the relationship between PaO2 (kPa) and PbtO2 (mmHg). | Throughout the duration of neuromonitoring in the neuro-ICU (1-30 days)
  Median goodness of fit (Pearsons R2)
Correlation between systemic lactate and microdialysis lactate when corrected for PbtO2 and cerebral perfusion pressure. | Throughout the duration of neuromonitoring in the neuro-ICU (1-30 days)
  Median goodness of fit (Pearsons R2)
The predictive value of glutamate measured by intracerebral microdialysis for episodes of neuroworsening | Throughout the duration of neuromonitoring in the neuro-ICU (1-30 days)
  Area under the curve
The predictive value of glutamate measured by intracerebral microdialysis for 6-month functional outcome | Throughout the duration of neuromonitoring in the neuro-ICU (1-30 days)
  Modified Rankin Scale

SECONDARY OUTCOMES:
Length of hospital stay | From admission until discharge (1-300 days)
  Time in days
Mixed effects linear regression of the relationship betwen PaO2 (kPa) and PbtO2 (mmHg). | Six months after admission to the neuro-ICU
  mmHg/kPa
Functional outcome at six months | Six months after admission to the neuro-ICU
  Modified Rankin Scale
Mortality at six months | Six months after admission to the neuro-ICU
  Percent
Length of stay in the ICU | From admission until discharge from the ICU (1-300 days)
  Time in days

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten W Møller, Study Chair — Rigshospitalet, Afdeling for bedøvelse og intensiv behandling
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fenger AW, Lund A, Vassilieva A, Andreasen TH, Ebdrup SR, Bodilsen TS, Jensen HR, Olsen MH, Moller K. Relationship Between Systemic and Cerebral Microdialysate Glucose in Patients With Severe Acute Brain Injury-A Retrospective Study. Acta Anaesthesiol Scand. 2025 Jul;69(6):e70078. doi: 10.1111/aas.70078. PMID 40528433